CLINICAL TRIAL: NCT07203508
Title: Effect of Tongue-to-Palate Resistance Training on Penetration-Aspiration Scale and Suprahyoid Muscle Electrical Activity in Geriatric Patients With Oropharyngeal Dysphagia
Brief Title: Effect of Tongue-to-Palate Resistance Training in Geriatric Patients With Oropharyngeal Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Melinda Harini, Dr. dr. Melinda Harini, Sp.K.F.R., Ger. (K), Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KET-1415/UN2.F1/ETIK/PPM.00.02
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Oropharyngeal Dysphagia; Geriatric Patients
Keywords: Rehabilitation; aspiration; dysphagia; swallowing; tongue
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: This study utilized a parallel-group design, which is the standard model for a two-arm randomized controlled trial (RCT). Participants were randomly allocated to one of two distinct intervention groups that proceeded concurrently throughout the trial duration. One group received the experimental Tongue-to-Palate Resistance Training (TPRT) intervention, while the parallel comparator group received an active control treatment consisting of standard dysphagia therapy. The outcomes for both groups were assessed and compared at identical time points (baseline, week 4, and week 8) to evaluate the relative efficacy of the TPRT intervention against the control condition.
Who Masked: Outcomes Assessor
Masking Description: While the participants, care providers, and investigators involved in delivering the interventions were not masked due to the nature of the exercise-based interventions, the study maintained a single-blind design. The key masked party was the outcomes assessor. Specifically, the rehabilitation medicine physician who performed the surface electromyography (sEMG) measurements and the radiologist and rehabilitation medicine specialist who analyzed the videofluoroscopic swallowing study (VFSS) recordings were blinded to group allocation. This was implemented to ensure objective and unbiased assessment of the primary outcome measures (suprahyoid muscle electrical activity and Penetration-Aspiration Scale scores)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tongue-to-Palate Resistance Training (TPRT) (Experimental): Participants in this arm performed a home-based Tongue-to-Palate Resistance Training (TPRT) program. The intervention consisted of pressing the tongue against the palate for 30 repetitions per session, five sessions per week, for a total of eight weeks. Participants were provided with video guidance and a logbook to record adherence, and were supported by a caregiver. This was a simple, device-free exercise regimen designed to strengthen the oropharyngeal and suprahyoid musculature.
  Interventions: Other: Tongue-to-Palate Resistance Training
- Standard Dysphagia Therapy (Active Comparator): Participants in this arm received the standard of care for oropharyngeal dysphagia. This included supervised, hospital-based sessions twice a week consisting of either Neuromuscular Electrical Stimulation (NMES) applied to the submental region or biofeedback swallowing therapy. Additionally, they were instructed to perform unsupervised Chin Tuck Against Resistance (CTAR) exercises at home. This arm represents the conventional, multi-modal rehabilitation approach against which the experimental TPRT intervention was compared.
  Interventions: Combination Product: Standard Dysphagia Therapy

INTERVENTIONS:
Other: Tongue-to-Palate Resistance Training — The Tongue-to-Palate Resistance Training (TPRT) is a home-based, device-free exercise program. Participants were instructed to press their tongue firmly against their hard palate and hold the contraction. The protocol consisted of 30 repetitions per session, performed five days a week for a duration of eight weeks. Adherence was supported through instructional videos, a caregiver, and a training logbook. The goal of the intervention is to strengthen the intrinsic and extrinsic tongue muscles and the suprahyoid muscle group to improve swallowing function.
  Other Names: Tongue Press Exercise; Tongue Strength Training
  Arms: Tongue-to-Palate Resistance Training (TPRT)
Combination Product: Standard Dysphagia Therapy — The active comparator consists of a conventional, multi-modal standard of care for oropharyngeal dysphagia. It includes in-clinic sessions twice a week featuring either Neuromuscular Electrical Stimulation (NMES), where electrodes are placed in the submental region to stimulate the swallowing muscles, or biofeedback swallowing therapy. Additionally, participants perform unsupervised Chin Tuck Against Resistance (CTAR) exercises at home. This arm represents the established clinical rehabilitation approach against which the experimental TPRT intervention is compared
  Other Names: Active Comparator; Conventional Dysphagia Therapy
  Arms: Standard Dysphagia Therapy

SUMMARY:
The goal of this randomized controlled trial is to learn if a home-based Tongue-to-Palate Resistance Training (TPRT) program can improve swallowing muscle activity and swallowing safety in geriatric patients (aged >60 years) with oropharyngeal dysphagia. The main questions it aims to answer are:

1. Does TPRT increase the electrical activity of the suprahyoid muscles (a key muscle group for swallowing) more than standard care?
2. Does TPRT reduce scores on the Penetration-Aspiration Scale (PAS), a measure of swallowing safety, more than standard care?
3. Researchers will compare the TPRT intervention group to the active control group to see if the simple, home-based TPRT exercise is as effective or more effective than standard hospital-based therapies.

Participants in the intervention group will:

Perform the TPRT exercise (pressing their tongue against the palate) for 30 repetitions, 5 times a week, for 8 weeks at home.

Be supported by a caregiver and use a video guide and logbook.

Participants in the control group will:

Receive standard hospital-based therapy twice a week, which may include Neuromuscular Electrical Stimulation (NMES) or biofeedback.

Perform unsupervised Chin Tuck Against Resistance (CTAR) exercises at home.

All participants will also receive education on safe swallowing techniques.

DETAILED DESCRIPTION:
Title: Effect of Tongue-to-Palate Resistance Training on Penetration-Aspiration Scale and Suprahyoid Muscle Electrical Activity in Geriatric Patients with Oropharyngeal Dysphagia: A Randomized Control Trial

Journal & Type: This is a manuscript for publication, presenting the results of a single-blind, randomized controlled trial (RCT).

Authors: The team is multi-disciplinary, consisting of experts in Internal Medicine, Physical Medicine and Rehabilitation (PM&R), and Radiology from Cipto Mangunkusumo Hospital/University of Indonesia, and a collaborator from Germany.

Background & Rationale:

Problem: Oropharyngeal dysphagia (difficulty swallowing) is a very common and serious problem in the elderly, leading to malnutrition, pneumonia from aspiration, and increased death rates.

Current Solutions: Existing therapies (like Shaker exercises or electrical stimulation) can be difficult for frail elderly patients to perform or require clinic visits.

Proposed Solution: Tongue-to-Palate Resistance Training (TPRT) is a simple, home-based exercise that could strengthen tongue and throat muscles, potentially improving swallowing. Preliminary studies showed it increases muscle activity, but robust evidence in geriatric patients was needed.

Objective: To determine if an 8-week home-based TPRT program is effective at improving swallowing muscle activity (measured by electromyography/sEMG) and swallowing safety (measured by the Penetration-Aspiration Scale on videofluoroscopy) in elderly dysphagia patients.

Methods:

Design: Single-blind Randomized Controlled Trial (RCT).

Participants: 20 elderly patients (>60 years) with confirmed oropharyngeal dysphagia. They had to have low baseline muscle activity and an available caregiver.

Intervention Group (n=9): Performed home-based TPRT (30 reps, 5x/week for 8 weeks) with video guidance and logbook monitoring.

Control Group (n=8): Received standard care, which included clinic-based Neuromuscular Electrical Stimulation (NMES) or biofeedback twice a week plus unsupervised home exercises (Chin Tuck Against Resistance).

Measurements:

Primary Outcome 1: Suprahyoid Muscle Activity. Measured using surface electromyography (sEMG) at baseline, 4 weeks, and 8 weeks.

Primary Outcome 2: Swallowing Safety. Measured using the Penetration-Aspiration Scale (PAS) via Videofluoroscopic Swallowing Study (VFSS) at baseline and 8 weeks.

Secondary Outcomes: Hyoid bone movement (crucial for swallowing) and Pharyngeal Transit Time (PTT) were also measured from the VFSS.

Analysis: Used advanced statistical tests (Repeated Measures ANOVA, Wilcoxon tests) to compare changes within and between groups over time.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years with a diagnosis of oropharyngeal dysphagia based on history, physical examination, and Videofluoroscopic Swallowing Study (VFSS)
* Initial measurement of suprahyoid muscle electrical activity ≤ 37.1 µV RMS
* Has not undergone any other swallowing exercises or is not currently participating in any swallowing exercise program within the past 2 weeks.
* Cooperative and willing to participate in the study by signing the informed consent form after receiving an explanation
* Has a caregiver who is willing to participate and is cooperative to ensure the patient follows the exercise protocol according to the study.

Exclusion Criteria:

* Cognitive impairment in the domains of memory, attention, or language based on the Montreal Cognitive Assessment - Indonesian version (MoCA-Ina), which would prevent the subject from following exercise instructions.
* Presence of other conditions causing dysphagia, such as oral cavity malignancy, history of radical neck dissection, or history of chemoradiotherapy to the neck region less than 3 months after the last session.
* Complete inability to move the tongue or initial suprahyoid muscle electrical activity measurement = 0 µV.
* Allergy to barium, potato starch, corn starch, xanthan gum, dairy products, or latex.
* Use of a pacemaker.

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Change in Penetration-Aspiration Scale (PAS) Score | Baseline and Week 8
  Change in swallowing safety as measured by the Penetration-Aspiration Scale (PAS). The PAS is an 8-point ordinal scale. The minimum score is 1 (no airway invasion) and the maximum score is 8 (aspiration of material into the airway with no reflexive response). A lower score on the PAS indicates a safer swallow and is a better outcome.
Change in Suprahyoid Muscle Electrical Activity | Baseline, Week 4, and Week 8
  The change in the electrical activity of the suprahyoid muscles (measured in microvolts root mean square, μV RMS) during a tongue press task and a dry swallow task. Measured using surface electromyography (sEMG).

SECONDARY OUTCOMES:
Change in Anterior Hyoid Excursion | Baseline and Week 8
  The change in the distance of forward (anterior) movement of the hyoid bone during swallowing, expressed as a percentage of the C2-C4 vertebral distance. Measured from VFSS.
Change in Superior Hyoid Excursion | Baseline and Week 8
  The change in the distance of upward (superior) movement of the hyoid bone during swallowing, expressed as a percentage of the C2-C4 vertebral distance. Measured from VFSS.
Change in Pharyngeal Transit Time (PTT) | Baseline and Week 8
  The change in the time (in seconds) taken for the bolus to travel from the point where the bolus tail passes the ramus of the mandible to when it passes through the upper esophageal sphincter. Measured from VFSS.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant confidentiality

REFERENCES:
- [Result] Zhang Z, Perera S, Donohue C, Kurosu A, Mahoney AS, Coyle JL, Sejdic E. The Prediction of Risk of Penetration-Aspiration Via Hyoid Bone Displacement Features. Dysphagia. 2020 Feb;35(1):66-72. doi: 10.1007/s00455-019-10000-5. Epub 2019 Mar 27. PMID 30919104
- [Result] Bingjie L, Tong Z, Xinting S, Jianmin X, Guijun J. Quantitative videofluoroscopic analysis of penetration-aspiration in post-stroke patients. Neurol India. 2010 Jan-Feb;58(1):42-7. doi: 10.4103/0028-3886.60395. PMID 20228462
- [Result] Kim H, Kown Y, Choi H. Home Based Dysphagia Rehabilitation for Stroke Patients Using Information and Communication Technology. J Int Acad Phys Ther Res. 2021;12(1):2267-71
- [Result] Pearson WG Jr, Hindson DF, Langmore SE, Zumwalt AC. Evaluating swallowing muscles essential for hyolaryngeal elevation by using muscle functional magnetic resonance imaging. Int J Radiat Oncol Biol Phys. 2013 Mar 1;85(3):735-40. doi: 10.1016/j.ijrobp.2012.07.2370. Epub 2012 Sep 18. PMID 22995662
- [Result] Han H, Shin G, Jun A, Park T, Ko D, Choi E, Kim Y. The Relation Between the Presence of Aspiration or Penetration and the Clinical Indicators of Dysphagia in Poststroke Survivors. Ann Rehabil Med. 2016 Feb;40(1):88-94. doi: 10.5535/arm.2016.40.1.88. Epub 2016 Feb 26. PMID 26949674
- [Result] Steele CM, Bailey GL, Chau T, Molfenter SM, Oshalla M, Waito AA, Zoratto DC. The relationship between hyoid and laryngeal displacement and swallowing impairment. Clin Otolaryngol. 2011 Feb;36(1):30-6. doi: 10.1111/j.1749-4486.2010.02219.x. PMID 21414151
- [Result] Hughes TD. The Effect of Two Rehabilitation Exercise on Submental Hyolaringeal Muscular Activity. Texas Christian University; 2015
- [Result] Steele CM, Bayley MT, Peladeau-Pigeon M, Nagy A, Namasivayam AM, Stokely SL, Wolkin T. A Randomized Trial Comparing Two Tongue-Pressure Resistance Training Protocols for Post-Stroke Dysphagia. Dysphagia. 2016 Jun;31(3):452-61. doi: 10.1007/s00455-016-9699-5. Epub 2016 Mar 2. PMID 26936446
- [Result] Rogus-Pulia N, Rusche N, Hind JA, Zielinski J, Gangnon R, Safdar N, Robbins J. Effects of Device-Facilitated Isometric Progressive Resistance Oropharyngeal Therapy on Swallowing and Health-Related Outcomes in Older Adults with Dysphagia. J Am Geriatr Soc. 2016 Feb;64(2):417-24. doi: 10.1111/jgs.13933. Epub 2016 Jan 25. PMID 26804715
- [Result] Oommen ER. Effects of Three Lingual Conditions on Submental Muscle Activity in Healthy Young and Old Adults. Ohio University; 2013
- [Result] Vaiman M, Eviatar E, Segal S. Surface electromyographic studies of swallowing in normal subjects: a review of 440 adults. Report 2. Quantitative data: amplitude measures. Otolaryngol Head Neck Surg. 2004 Nov;131(5):773-80. doi: 10.1016/j.otohns.2004.03.014. PMID 15523465
- [Result] Furlan R et al. Comparison of the electric activity of the suprahyoid muscles during different lingual exercises. Audiol Commun. 2015;20(3):203-9
- [Result] Gutierrez DL. A Comparison of Two Devices for Isometric Lingual Strengthening in Healthy Adults A COMPARISON OF TWO DEVICES FOR ISOMETRIC. 2020
- [Result] Palmer PM, Jaffe DM, McCulloch TM, Finnegan EM, Van Daele DJ, Luschei ES. Quantitative contributions of the muscles of the tongue, floor-of-mouth, jaw, and velum to tongue-to-palate pressure generation. J Speech Lang Hear Res. 2008 Aug;51(4):828-35. doi: 10.1044/1092-4388(2008/060). PMID 18658054
- [Result] Park JS, Kim HJ, Oh DH. Effect of tongue strength training using the Iowa Oral Performance Instrument in stroke patients with dysphagia. J Phys Ther Sci. 2015 Dec;27(12):3631-4. doi: 10.1589/jpts.27.3631. Epub 2015 Dec 28. PMID 26834320
- [Result] Robbins J, Kays SA, Gangnon RE, Hind JA, Hewitt AL, Gentry LR, Taylor AJ. The effects of lingual exercise in stroke patients with dysphagia. Arch Phys Med Rehabil. 2007 Feb;88(2):150-8. doi: 10.1016/j.apmr.2006.11.002. PMID 17270511
- [Result] Robbins J, Gangnon RE, Theis SM, Kays SA, Hewitt AL, Hind JA. The effects of lingual exercise on swallowing in older adults. J Am Geriatr Soc. 2005 Sep;53(9):1483-9. doi: 10.1111/j.1532-5415.2005.53467.x. PMID 16137276
- [Result] Gabriel DA, Kamen G, Frost G. Neural adaptations to resistive exercise: mechanisms and recommendations for training practices. Sports Med. 2006;36(2):133-49. doi: 10.2165/00007256-200636020-00004. PMID 16464122
- [Result] Lavin KM, Roberts BM, Fry CS, Moro T, Rasmussen BB, Bamman MM. The Importance of Resistance Exercise Training to Combat Neuromuscular Aging. Physiology (Bethesda). 2019 Mar 1;34(2):112-122. doi: 10.1152/physiol.00044.2018. PMID 30724133
- [Result] Salles B De, Simão R, Fleck S. Effects of Resistance Training on older adults. Sports Medicine. 2010;34(5):441-50
- [Result] Plaza E, Ruviaro Busanello-Stella A. Effects of a tongue training program in Parkinson's disease: Analysis of electrical activity and strength of suprahyoid muscles. J Electromyogr Kinesiol. 2022 Apr;63:102642. doi: 10.1016/j.jelekin.2022.102642. Epub 2022 Feb 12. PMID 35189571
- [Result] Park JS, Lee SH, Jung SH, Choi JB, Jung YJ. Tongue strengthening exercise is effective in improving the oropharyngeal muscles associated with swallowing in community-dwelling older adults in South Korea: A randomized trial. Medicine (Baltimore). 2019 Oct;98(40):e17304. doi: 10.1097/MD.0000000000017304. PMID 31577721
- [Result] Vaiman M. Standardization of surface electromyography utilized to evaluate patients with dysphagia. Head Face Med. 2007 Jun 6;3:26. doi: 10.1186/1746-160X-3-26. PMID 17553152
- [Result] Yoshida M, Groher ME, Crary MA, Mann GC, Akagawa Y. Comparison of surface electromyographic (sEMG) activity of submental muscles between the head lift and tongue press exercises as a therapeutic exercise for pharyngeal dysphagia. Gerodontology. 2007 Jun;24(2):111-6. doi: 10.1111/j.1741-2358.2007.00164.x. PMID 17518959
- [Result] Palmer PM, Luschei ES, Jaffe D, McCulloch TM. Contributions of individual muscles to the submental surface electromyogram during swallowing. J Speech Lang Hear Res. 1999 Dec;42(6):1378-91. doi: 10.1044/jslhr.4206.1378. PMID 10599620
- [Result] Wirth R, Dziewas R, Beck AM, Clave P, Hamdy S, Heppner HJ, Langmore S, Leischker AH, Martino R, Pluschinski P, Rosler A, Shaker R, Warnecke T, Sieber CC, Volkert D. Oropharyngeal dysphagia in older persons - from pathophysiology to adequate intervention: a review and summary of an international expert meeting. Clin Interv Aging. 2016 Feb 23;11:189-208. doi: 10.2147/CIA.S97481. eCollection 2016. PMID 26966356
- [Result] Reis VS dos, Araújo TG de, Furlan RMMM, Motta AR. Correlation between tongue pressure and electrical activity of the suprahyoid muscles. Revista CEFAC. 2017;19(6):792-800
- [Result] Harini M, Nathania E. The Effectiveness of Tongue Palatal Resistance Training on Increasing Suprahyoid Muscle Strength in Patients with Oropharyngeal Dysphagia: A Home Exercise Program during the Covid-19 Pandemic. ASEAN Journal of Rehabilitation Medicine. 2021;32(Fourthcoming):41-3
- [Result] Lee KH, Jung ES, Choi YY. Effects of lingual exercises on oral muscle strength and salivary flow rate in elderly adults: a randomized clinical trial. Geriatr Gerontol Int. 2020 Jul;20(7):697-703. doi: 10.1111/ggi.13944. Epub 2020 Jun 2. PMID 32489001
- [Result] Namiki C, Hara K, Tohara H, Kobayashi K, Chantaramanee A, Nakagawa K, Saitou T, Yamaguchi K, Yoshimi K, Nakane A, Minakuchi S. Tongue-pressure resistance training improves tongue and suprahyoid muscle functions simultaneously. Clin Interv Aging. 2019 Mar 22;14:601-608. doi: 10.2147/CIA.S194808. eCollection 2019. PMID 30962680
- [Result] Kim HD, Choi JB, Yoo SJ, Chang MY, Lee SW, Park JS. Tongue-to-palate resistance training improves tongue strength and oropharyngeal swallowing function in subacute stroke survivors with dysphagia. J Oral Rehabil. 2017 Jan;44(1):59-64. doi: 10.1111/joor.12461. PMID 27883209
- [Result] Park JS, Hwang NK, Kim HH, Choi JB, Chang MY, Jung YJ. Effects of lingual strength training on oropharyngeal muscles in South Korean adults. J Oral Rehabil. 2019 Nov;46(11):1036-1041. doi: 10.1111/joor.12835. Epub 2019 Jul 2. PMID 31206763
- [Result] Park T. Effects of Oropharyngeal Strengthening Exercise (OSE) on Tongue Strength, Submental Muscle Activity, and Quality of Life in a Healthy Elderly Population. Ohio University; 2015
- [Result] Yano J, Yamamoto-Shimizu S, Yokoyama T, Kumakura I, Hanayama K, Tsubahara A. Effects of Tongue-Strengthening Exercise on the Geniohyoid Muscle in Young Healthy Adults. Dysphagia. 2020 Feb;35(1):110-116. doi: 10.1007/s00455-019-10011-2. Epub 2019 Apr 22. PMID 31011804
- [Result] Smithard DG. Dysphagia : A Geriatric Giant ? The Normal Swallow. iMedPub Journals. 2016;2(1:5):1-7
- [Result] Penalva-Arigita A, Prats R, Lecha M, Sansano A, Vila L. Prevalence of dysphagia in a regional hospital setting: Acute care hospital and a geriatric sociosanitary care hospital: A cross-sectional study. Clin Nutr ESPEN. 2019 Oct;33:86-90. doi: 10.1016/j.clnesp.2019.07.003. Epub 2019 Jul 24. PMID 31451280
- [Result] Baijens LW, Clave P, Cras P, Ekberg O, Forster A, Kolb GF, Leners JC, Masiero S, Mateos-Nozal J, Ortega O, Smithard DG, Speyer R, Walshe M. European Society for Swallowing Disorders - European Union Geriatric Medicine Society white paper: oropharyngeal dysphagia as a geriatric syndrome. Clin Interv Aging. 2016 Oct 7;11:1403-1428. doi: 10.2147/CIA.S107750. eCollection 2016. PMID 27785002
- [Result] Clave P, Shaker R. Dysphagia: current reality and scope of the problem. Nat Rev Gastroenterol Hepatol. 2015 May;12(5):259-70. doi: 10.1038/nrgastro.2015.49. Epub 2015 Apr 7. PMID 25850008
- [Result] Clave P, Rofes L, Carrion S, Ortega O, Cabre M, Serra-Prat M, Arreola V. Pathophysiology, relevance and natural history of oropharyngeal dysphagia among older people. Nestle Nutr Inst Workshop Ser. 2012;72:57-66. doi: 10.1159/000339986. Epub 2012 Sep 24. PMID 23052001
- [Result] Rofes L, Arreola V, Almirall J, Cabre M, Campins L, Garcia-Peris P, Speyer R, Clave P. Diagnosis and management of oropharyngeal Dysphagia and its nutritional and respiratory complications in the elderly. Gastroenterol Res Pract. 2011;2011:818979. doi: 10.1155/2011/818979. Epub 2010 Aug 3. PMID 20811545

DOCUMENTS (2):
  • Study Protocol (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT07203508/Prot_000.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT07203508/ICF_001.pdf